CLINICAL TRIAL: NCT04369820
Title: C5a Receptor Expression in Circulating Myeloid Cells in ARDS Secondary to COVID-19
Brief Title: C5a Receptor Expression - COVID-19 (C5-COV)
Acronym: C5-COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-14; IDRCB (Other: 2020-A00757-32)
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19; ARDS; C5a receptors
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 PATIENTS (Experimental): Two blood samples (40mL) at 2 different points in time:
  1. Within the first 72 hours of medical care in resuscitation unit or department.
  2. Between the 5th and the 10th day of medical care (ideally at the end of the first week) or on the day of discharge of patient if it is earlier, or of death if it takes place earlier.
  Interventions: Other: draw blood

INTERVENTIONS:
Other: draw blood — 40 mL blood sample will be taken within the first three days of hospitalization, a second sample will be taken between the 5th and 10th day of hospitalization and a third sample will be taken on the 10th day of hospitalization or the day of discharge if earlier.

SUMMARY:
The pathophysiology of ARDS is linked to an uncontrolled inflammatory response at the level of alveolo-capillary membrane, mediated by neutrophils and mononuclear cells. The complement system and anaphylatoxin C5a have shown central role in the recruitment of these pro-inflammatory cells and more broadly in the genesis of cytokinic storm syndrome. C5a acts via receptors C5aR and C5L2.

This is a preliminary study aimed at studying the expression of the C5a receptor on myeloid cells in peripheral blood of patients with ARDS secondary to COVID-19.

This study has of primary objective to show there is an overexpression of the C5a receptor in patients with ARDS secondary to COVID-19 compared to control patients (patients with COVID-19 without respiratory distress and healthy volunteers).

The medium-term objective is to develop a clinical trial to test the effectiveness of anti-C5aR antibody in this condition.

DETAILED DESCRIPTION:
The pathophysiology of ARDS is linked to an uncontrolled inflammatory response at the level of alveolo-capillary membrane, mediated by neutrophils and mononuclear cells. The complement system and anaphylatoxin C5a have shown central role in the recruitment of these pro-inflammatory cells and more broadly in the genesis of cytokinic storm syndrome. C5a acts via receptors C5aR and C5L2.

This is a preliminary study aimed at studying the expression of the C5a receptor on myeloid cells in peripheral blood of patients with ARDS secondary to COVID-19.

This study has of primary objective to show there is an overexpression of the C5a receptor in patients with ARDS secondary to COVID-19 compared to control patients (patients with COVID-19 without respiratory distress and healthy volunteers).

The medium-term objective is to develop a clinical trial to test the effectiveness of anti-C5aR antibody in this condition.

ELIGIBILITY:
Inclusion Criteria:

For patients in resuscitation unit with ARDS linked to COVID-19:

* Patient under invasive mechanical ventilation
* PaO2 / FiO2 <300
* PCR SARS-CoV-2 positive in a pharyngeal or respiratory sample

For control patients with COVID-19 without ARDS

* Oxygen flow always less than 5 L / min
* PCR SARS-CoV-2 positive in a pharyngeal or respiratory sample
* No passage in resuscitation unit
* Favorable evolution

Exclusion Criteria:

* Minors
* Patient deprived of liberty
* Patient's refusal to participate at study
* Patient for whom therapeutic limitation measures such as non-admission to intensive care have been issued
* Medullar aplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Show an overexpression of C5a receptor in patients with ARDS secondary to COVID-19 compared to control patients (patients with COVID-19 without respiratory distress and healthy volunteers). | 72 hours
  The endpoint is the expression of the C5a receptor (C5aR) in peripheral blood myeloid cells, expressed as a percentage of cells expressing C5a receptor and as median fluorescence intensity (MFI), during the first 72 hours of patient management in resuscitation unit.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie EGP GARRIDO-PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Background] Kinross P, Suetens C, Dias JG, Alexakis L, Wijermans A, Colzani E, Monnet DL; European Centre for Disease Prevention and Control (ECDC) Public Health Emergency Team; ECDC Public Health Emergency Team. Rapidly increasing cumulative incidence of coronavirus disease (COVID-19) in the European Union/European Economic Area and the United Kingdom, 1 January to 15 March 2020. Euro Surveill. 2020 Mar;25(11):2000285. doi: 10.2807/1560-7917.ES.2020.25.11.2000285. Epub 2020 Mar 16. PMID 32186277
- [Background] Parmet WE, Sinha MS. Covid-19 - The Law and Limits of Quarantine. N Engl J Med. 2020 Apr 9;382(15):e28. doi: 10.1056/NEJMp2004211. Epub 2020 Mar 18. No abstract available. PMID 32187460
- [Background] Gostin LO, Hodge JG Jr, Wiley LF. Presidential Powers and Response to COVID-19. JAMA. 2020 Apr 28;323(16):1547-1548. doi: 10.1001/jama.2020.4335. No abstract available. PMID 32186661
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Herrero R, Sanchez G, Lorente JA. New insights into the mechanisms of pulmonary edema in acute lung injury. Ann Transl Med. 2018 Jan;6(2):32. doi: 10.21037/atm.2017.12.18. PMID 29430449
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Gralinski LE, Sheahan TP, Morrison TE, Menachery VD, Jensen K, Leist SR, Whitmore A, Heise MT, Baric RS. Complement Activation Contributes to Severe Acute Respiratory Syndrome Coronavirus Pathogenesis. mBio. 2018 Oct 9;9(5):e01753-18. doi: 10.1128/mBio.01753-18. PMID 30301856
- [Background] Wang R, Xiao H, Guo R, Li Y, Shen B. The role of C5a in acute lung injury induced by highly pathogenic viral infections. Emerg Microbes Infect. 2015 May;4(5):e28. doi: 10.1038/emi.2015.28. Epub 2015 May 6. PMID 26060601
- [Background] Jiang Y, Zhao G, Song N, Li P, Chen Y, Guo Y, Li J, Du L, Jiang S, Guo R, Sun S, Zhou Y. Blockade of the C5a-C5aR axis alleviates lung damage in hDPP4-transgenic mice infected with MERS-CoV. Emerg Microbes Infect. 2018 Apr 24;7(1):77. doi: 10.1038/s41426-018-0063-8. PMID 29691378
- [Background] Stevens JH, O'Hanley P, Shapiro JM, Mihm FG, Satoh PS, Collins JA, Raffin TA. Effects of anti-C5a antibodies on the adult respiratory distress syndrome in septic primates. J Clin Invest. 1986 Jun;77(6):1812-6. doi: 10.1172/JCI112506. PMID 3711336
- [Background] Czermak BJ, Sarma V, Pierson CL, Warner RL, Huber-Lang M, Bless NM, Schmal H, Friedl HP, Ward PA. Protective effects of C5a blockade in sepsis. Nat Med. 1999 Jul;5(7):788-92. doi: 10.1038/10512. PMID 10395324